Title: One Key Question, Pilot Study Phase II

Study EH#: 18-343

NCT03947788

January 23, 2018

## Appendix D: Oral recruitment and consent script

Hi, my name is [insert name] and I work for NorthShore. Would you be interested in participating in a short research survey today to help improve women's reproductive health?"

or

Hi, my name is [insert name] and I work for NorthShore. Would you be interested in participating in a short research survey today to help improve women's reproductive health?" This survey should take approximately 2 minutes.

Yes (continue with script)

No

Thank you for your time. Have a nice day.

The purpose of this study is to improve reproductive health care which means providing birth control and/or information about having a healthy pregnancy to women who want it. No identifying information will be collected about you for this research. No one will know your name or how you answered these questions. These surveys will not be part of your medical record. Your response to the survey questions will be used for research only. Your participation is optional. There will be no penalty or change in medical care for refusing to participate.

There are eligibility criteria for participating in this study. To identify if you are eligible I need to ask you one question. Are you a female between the ages of 18-49, currently not pregnant, and seeing your provider or a nurse practitioner today?

or

There are eligibility criteria for participating in this study. To identify if you are eligible I need to ask you a few questions.

Are you between the ages of 18-49 years old?

Are you pregnant?

Are you seeing your doctor or nurse practitioner today?

If participant does not meet one or all criteria...

Thank you for listening. Unfortunately you do not meet the criteria to participate.

If participant is eligible, continue with script

Thank you! You are eligible to continue. If you have any questions or concerns about the research study, please feel free to let me know and I can give you the contact information of our study's principal investigator.